CLINICAL TRIAL: NCT05451836
Title: Patient, Physician, and Organizational Factors Influencing Decision-making for Antibiotic Use, and N-of-1 Trials of Interventions to Improve the Decision-making
Brief Title: N-of-1 Trials of Interventions to Improve Decision-making for Antibiotic Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Changi General Hospital (Other); Khoo Teck Puat Hospital (Other); National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Chow Li Ping Angela, Head and Senior Consultant, Tan Tock Seng Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: NMRC/CSAINV18MAY0007/2019
Record Dates: First submitted 2022-07-03; First posted 2022-07-11 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Antimicrobial Resistance

STUDY DESIGN:
Intervention Model Description: Interrupted time series quasi-experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 (Two emergency departments) will receive patient education leaflets for 6 months and will receive physician feedback for the next 6 months on top of the patient education.
  Interventions: Other: Patient education leaflets; Other: Physician feedback
- Group 2 (Experimental): Group 1 (Two emergency departments) will receive physician feedback for 6 months and will receive patient education leaflets for the next 6 months on top of the physician feedback.
  Interventions: Other: Patient education leaflets; Other: Physician feedback

INTERVENTIONS:
Other: Patient education leaflets — Patients who attend the emergency department with upper respiratory tract infections will be provided with patient education leaflets on appropriate antibiotic use and antimicrobial resistance. The leaflets are available in the four national languages in Singapore.
Other: Physician feedback — All physicians working in the emergency department will receive a text message from their department head on their antibiotic prescribing rates every two months.

SUMMARY:
Antibiotics have brought about a substantial reduction in infectious mortality. However, inappropriate antibiotic use has driven the rapid increase in antibiotic resistance. The Centers for Disease Control and Prevention estimates that at least 2 million people in the United States (US) become infected with antibiotic-resistant bacteria each year, and at least 23,000 people die each year as a direct result of these infections.

Antimicrobial stewardship programs have largely focused on inpatient settings and have excluded emergency departments (ED). The ED is a unique healthcare setting which is distinct from inpatient and other ambulatory settings. Given the many factors that could influence inappropriate antibiotic prescribing, a one-size-fits-all approach is unlikely to work for all physicians and all regions. Hence, the design and implementation of tailored interventions based on the understanding of the local patient, physician, and ED organizational factors are pertinent for the interventions. The team has conducted a mixed-methods study to understand the patient, physician, and organisational factors that influence antibiotic prescribing in the local EDs. The findings of the study were used to design two interventions which will be implemented in four EDs in Singapore to reduce the inappropriate antibiotic prescribing in the ED.

This study aims to evaluate the effectiveness of 2 tailored antimicrobial stewardship interventions in reducing antibiotic prescribing rates for uncomplicated URTI patients attending four adult EDs in Singapore:

1. Patient education via information leaflets addressing knowledge-, perception-, and belief-gaps of the local patient population on antibiotic use for URTI
2. Two-monthly physician feedback on their antibiotic prescribing rates by senior ED doctors coupled with bite-sized information on good antibiotic prescribing practices.

The study will include an initial control period of 18 months where none of the 4 hospitals will be exposed to the interventions. At the beginning of the intervention period, the 4 hospitals will be randomly assigned to one of the 2 interventions (Patient education or physician feedback). At the end of 6 months, all hospitals will receive the other intervention and be exposed to both interventions concurrently. Data will be collected for another 6 months to assess if the effects of the interventions are persistent.

DETAILED DESCRIPTION:
Antibiotics, along with improved sanitation and vaccination, have brought about a substantial reduction in infectious mortality. However, inappropriate antibiotic use has driven the rapid increase in antibiotic resistance. The Centers for Disease Control and Prevention estimates that at least 2 million people in the United States (US) become infected with antibiotic-resistant bacteria each year, and at least 23,000 people die each year as a direct result of these infections.

To date, antimicrobial stewardship programs attempting to optimize antibiotic therapy and clinical outcomes have largely focused on inpatient settings and have excluded emergency departments (ED). The ED is a unique healthcare setting which is distinct from inpatient and other ambulatory settings. Given the multi-factorial nature of inappropriate antibiotic prescribing, it is unlikely that a single approach will work for all physicians in all regions. Hence, the design and implementation of tailored interventions based on the understanding of the local patient, physician, and ED organizational factors are pertinent for the interventions. The team has conducted a mixed-methods study to understand the patient, physician, and organisational factors that influence antibiotic prescribing in the local EDs. The findings of the study were used to design two interventions which will be implemented in four EDs in Singapore to reduce the inappropriate antibiotic prescribing in the ED.

This study aims to evaluate the effectiveness of 2 tailored antimicrobial stewardship interventions in reducing antibiotic prescribing rates for uncomplicated URTI patients attending four adult EDs in Singapore:

1. Patient education via information leaflets addressing knowledge-, perception-, and belief-gaps of the local patient population on antibiotic use for URTI
2. Two-monthly physician feedback on their antibiotic prescribing rates by senior ED doctors coupled with bite-sized information on good antibiotic prescribing practices.

Using the stepped wedge design, the study will include an initial control period of 18 months where none of the 4 hospitals will be exposed to the interventions. During the intervention period, the 4 hospitals will be randomly assigned to one of the 2 tailored interventions. At the end of 6 months, all hospitals will receive the other intervention and be exposed to both interventions concurrently. Data will be collected for another 6 months to assess the persistence of the effects of the interventions.

Patient educational materials: Education materials (patient leaflets) will be made available at the Emergency Departments of the participating sites. Patients will be exposed to these materials while visiting the Emergency Department prior to their consultation with the physician.

Feedback to individual physicians by senior doctors: Messages containing the individual antibiotic prescribing rate of each physician in the past month will be sent every two months to the respective physician by their department head (or senior doctor) via Tiger Text. The bite-sized information on tips to reduce antibiotic prescribing for URTI will be sent together with the personalised message.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Adults aged 21 years and above
* Attendance at any of the study sites' Emergency Department: National University Hospital, Khoo Teck Puat Hospital, Changi General Hospital and Tan Tock Seng Hospital
* Presenting with upper respiratory tract infections

Physicians:

* Working at any of the study sites' Emergency Department: National University Hospital (NUH), Khoo Teck Puat Hospital (KTPH), Changi General Hospital (CGH), Tan Tock Seng Hospital (TTSH) and Sengkang General Hospital (SKH), during the study period

Exclusion Criteria:

Nil

Ages: 21 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15157 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Antibiotic prescribing rates | Measured monthly for 15 months
  The antibiotic prescribing rates are computed by dividing the number of URTI patients prescribed with antibiotics with the total number of URTI seen by the physician. The data is obtained from the electronic medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Chow, Ph.D, Principal Investigator — Tan Tock Seng Hospital
Locations (4):
- Singapore (4):
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No
Only the site-PI will receive data on the antibiotic prescribing rates of the ED physicians for them to provide the physician feedback. The data of one site will not be shared with the site-PIs of other sites to preserve participant confidentiality.

REFERENCES:
- [Derived] Attal H, Huang Z, Kuan WS, Weng Y, Tan HY, Seow E, Peng LL, Lim HC, Chow A. N-of-1 Trials of Antimicrobial Stewardship Interventions to Optimize Antibiotic Prescribing for Upper Respiratory Tract Infection in Emergency Departments: Protocol for a Quasi-Experimental Study. JMIR Res Protoc. 2024 Feb 21;13:e50417. doi: 10.2196/50417. PMID 38381495